CLINICAL TRIAL: NCT07362186
Title: A Phase III, Open-Label, Multicenter, Randomized, Parallel-Group Study to Evaluate the Efficacy and Safety of LM-108 in Combination With Toripalimab Versus Paclitaxel Injection as Second-Line Therapy for CCR8-Positive Locally Advanced or Metastatic Gastric Cancer/Gastroesophageal Junction Adenocarcinoma
Brief Title: LM-108 in Combination With Toripalimab Versus Paclitaxel Injection for the Treatment of Subjects With CCR8-Positive Gastric and Gastroesophageal Junction Adenocarcinoma
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: LaNova Medicines Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LM108-03-202
Record Dates: First submitted 2026-01-07; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Locally Advanced or Metastatic GC and GCJ Adenocarcinoma
MeSH Terms: interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LM-108 in combination with Toripalimab (Experimental)
  Interventions: Drug: LM-108 in combination with Toripalimab
- Paclitaxel injection intravenous infusion (Active Comparator)
  Interventions: Drug: Paclitaxel injection intravenous infusion

INTERVENTIONS:
Drug: LM-108 in combination with Toripalimab — LM-108 combined with Toripalimab administered intravenously on Day 1 every 3 weeks
  Arms: LM-108 in combination with Toripalimab
Drug: Paclitaxel injection intravenous infusion — Paclitaxel injection administered at a dose of 80 mg/m² on Day 1, 8, and 15 every 4 weeks
  Arms: Paclitaxel injection intravenous infusion

SUMMARY:
This is a phase III， Multicenter, Randomized study， evaluating the efficacy and Safety of LM-108(an Anti-CCR8 mAb) in combination With Toripalimab Versus Paclitaxel Injection in subjects with CCR8-Positive locally advanced or metastatic Gastric Cancer and Gastroesophageal Junction Adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals who are willing to participate in the study and sign the informed consent form (ICF) prior to any procedure.
2. Age 18 years or older, male or female.
3. Weight ≥ 40 kg or Body Mass Index (BMI)≥ 18.5 kg/m²
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
5. Life expectancy ≥ 3 months.
6. Individuals must have histologically or cytologically confirmed locally advanced or metastatic gastric/gastroesophageal junction adenocarcinoma and be ineligible for curative surgery or radiotherapy.
7. Confirmed CCR8-positive by the central laboratory.
8. HER2-negative, low-expressing, or non-expressing.
9. Individuals must experience radiographic progression during or after prior standard first-line therapy, or who developed intolerance to treatment due to chemotherapy-related toxicity
10. At least one lesion.
11. Have appropriate organ and marrow function in laboratory examinations.
12. Women of childbearing potential have a negative pregnancy test and must not be breastfeeding. All of reproductive potential agree to use effective contraception throughout the study period and for 6 months after the last dose of study drug.

Exclusion Criteria:

1. Received treatment targeting the same target or other drugs acting on regulatory T cells (Tregs).
2. Received antitumor treatments such as chemotherapy, radiotherapy, biological therapy, immunotherapy, or Chinese herbal medicine or Chinese herbal preparations within 2-4 weeks (depending on the specific anticancer drug) prior to the first dose.
3. Received anti-PD-(L)1 antibody immunotherapy and experienced disease progression confirmed by RECIST 1.1 assessment within ≤2 months after treatment initiation.
4. Use of any live vaccine within 4 weeks prior to the first dosing of study drugs.
5. Individuals who received major surgery or interventional treatment within 4 weeks prior to the first dosing of study drugs.
6. Individuals who take systemic corticosteroids (> 10 mg daily prednisone equivalents) or other systemic immunosuppressive medications within 2 weeks prior to the first dosing of study drugs.
7. Any adverse event from prior anti-tumor therapy has not yet recovered to ≤ grade 1 of CTCAE v6.0, individuals who experienced ≥ Grade 3 immune-related adverse events during prior immunotherapy, or terminated prior immunotherapy due to severe or life-threatening immune-related adverse events.
8. Any other pathological type.
9. Uncontrollable clinical third-space fluid accumulation.
10. Unstable or progressive central nervous system (CNS) metastases or carcinomatous meningitis (meningeal metastases).
11. Individuals with a known history of autoimmune diseases.
12. For individuals with drug allergies or contraindications.
13. The investigator determined that there are other situations that are not suitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2026-04-03 (Estimated); Primary Completion 2028-08-17 (Estimated); Study Completion 2028-09-28 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | up to 42 months
  OS was defined as the time from date of randomization until death from any cause

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | up to 42 months
  PFS was defined as the time from date of randomization until first objective radiographic tumor progression or death from any cause, based on Investigator assessment
Objective response rate (ORR) | up to 42 months
  ORR is defined as the proportion of subjects achieving the best overall response (BOR) of CR or PR. BOR refers to the best response recorded during the period from the date of randomization to the date of objective progression documented according to RECIST 1.1 criteria or the date of initiation of subsequent antitumor therapy (whichever occurs first).
Duration of response (DOR) | Time from initial response (CR or PR) to date of documented disease progression or death (due to any cause) whichever occurs first, up to 42 months
  defined time from the initial response (CR or PR) until documented tumor progression or death from any cause and based on Investigator assessment.
Disease control rate (DCR) | From start of treatment to date of documented disease progression, up to approximately 42 months
  defined as the proportion of participants who achieved CR, PR, or stable disease (SD) , based on Investigator assessment.
Incidence of adverse events (AEs) | up to 42 months

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China